CLINICAL TRIAL: NCT01124071
Title: A 13 Week Study to Examine the Effectiveness of the Korean Diet on Weight, Blood Pressure, Metabolic Parameters and Disease Control in an Australian Overweight and Obese Population.
Brief Title: Korean Diet Efficacy Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sydney (Other)
Collaborators: Inje University (Other); Korea Agro-Fisheries Trade Corporation, Seoul, Korea (Unknown); Ministry for Food, Agriculture, Forestry and Fisheries, Korea (Other Government)
Responsible Party: Professor Ian Caterson, Boden Institute of Obesity, Nutrition & Exercise The University of Sydney
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 11-2009/12124
Record Dates: First submitted 2010-04-22; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-04

CONDITIONS: Obesity
Keywords: Korean Diet
MeSH Terms: conditions — Obesity | interventions — Diet, Western

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Korean Diet (Active Comparator): Provision of 2 Korean meals per day, 6 days per week
  Interventions: Behavioral: Provision of 2 Korean meals per day 6 days per week
- Western Diet (Active Comparator): Lifestyle counseling, dietary advice, grocery vouchers
  Interventions: Behavioral: Western Diet

INTERVENTIONS:
Behavioral: Provision of 2 Korean meals per day 6 days per week — At each participant's baseline visit, participant's will have an individualised lifestyle session addressing dietary and exercise goals and techniques to achieve weight loss. Participants in the Korean diet group will pick up lunch and evening meals Monday-Friday. Raw ingredients and cooking instructions will also be provided on friday for saturday meal preparation. Ongoing lifestyle sessions will be performed weekly for participants.
  Arms: Korean Diet
Behavioral: Western Diet — At each participant's baseline visit, participant's will have an individualised lifestyle session addressing dietary and exercise goals and techniques to achieve weight loss. Participants in the Western diet group will be provided with a Western recipe cookbook and food vouchers (weekly) to purchase the necessary ingredients for the Western meal preparation. Ongoing lifestyle sessions will be performed weekly for participants.
  Arms: Western Diet

SUMMARY:
To determine:

1. the acceptability of a Korean diet to an Australian overweight and obese population
2. which Korean recipes are easily prepared
3. the effect of a Korean diet on weight, blood pressure, and metabolic complications of obesity in this population.

DETAILED DESCRIPTION:
The primary endpoint (Korean diet acceptability) will be assessed by reliability tested questionnaire, dietary compliance, and quantities of food returned over the 12 weeks.

Analysis of differences in weight loss will be based on all participants with a baseline and a 12-week weight assessment. In order to investigate the impact of missing data, all subjects will be analysed using last weight observation carried forward and baseline weight carried forward.

Other secondary endpoints will determine the effect of the Korean diet on blood pressure, metabolic parameters and chronic metabolic disease control in the Australian population.

ELIGIBILITY:
Inclusion Criteria:

* Residents of metropolitan Sydney
* Aged 18-65 years
* BMI 25-45kg/m2

Exclusion Criteria:

* Diabetes treated with oral medications or insulin
* Unstable angina or recent onset of cardiovascular disease
* Serious hepatic or renal disease
* serum transaminases (ALT or AST) > 2.5 times upper limit of normal
* serum creatinine > 1.5 times upper limit of normal or urinary microalbumin >40 mg/L or eGFR < 60ml/min/1.73m²
* Alcohol or illicit drug abuse
* Pregnant, breastfeeding, or planning pregnancy during the study
* Serious gastrointestinal disease (inflammatory bowel disease, active peptic ulcer, recent helicobacter pylori treatment)
* Treatment for an eating disorder, weight loss medications and other drugs that affect body weight e.g. some anti-psychotics, anti-depressants, or corticosteroids
* Hypothyroidism defined by elevated thyroid stimulating hormone (TSH) and low free thyroxine (fT4), or current hyperthyroidism under treatment
* Participation in another weight loss clinical trial within past 3 months
* Individuals who have lost >10% weight within past 3 months
* Vegetarian eating practices
* Inability to cook or lack of facilities for home cooking
* Inability to read and write English
* Subjects who frequently change smoking habits or who have stopped smoking within 6 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
1. To investigate the acceptability of a Korean diet in overweight and obese Australians. | 13 weeks
  This will be determined at baseline and 4 week timepoints throughout the study by participants completing a Food Acceptability Questionnaire (FAQ). The FAQ addresses 10 components of food acceptability along a 7-point Likeart scale. The FAQ is a recognised instrument for testing food acceptability.
2. To examine the differences in weight loss between the Korean diet intervention and the Western diet intervention in overweight and obese Australians. | 13 weeks
  This will be determined by assessing differences at baseline and 12 weeks for weight, BMI and percent BMI change.

SECONDARY OUTCOMES:
To investigate changes in a number of indicators of metabolic disease in both groups - including anthropometry, Blood Glucose Levels, insulin sensitivity, lipid profiles, liver function, hormone function and inflammatory markers. | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ian D Caterson, AM, MBBS, BSc(Med), PhD, FRACP, Principal Investigator — University of Sydney
Locations (1):
- The University of Sydney, Sydney, New South Wales, Australia